CLINICAL TRIAL: NCT00983125
Title: Effects of a Systematic Addition of Clonidine in the Local Anaesthetic and Opiate Solution for Epidural Patient Controlled Analgesia in Labour (Levobupivacaine 0.568 mg.mLl-1 + Sufentanil 0.45 µg.mL-1)
Brief Title: Systematic Clonidine for Epidural Analgesia in Labour
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0058
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Labour
Keywords: Labour; Epidural analgesia; Clonidine; Levobupivacaine; Opiates; Patient-controlled; Active spontaneous labour requiring epidural analgesia
MeSH Terms: interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- clonidine (Experimental)
  Interventions: Drug: Clonidine
- no clonidine (Other)
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — Addition of a non-labeled drug (clonidine) in one of the two arm of the study, with randomisation.
  To compare the effects of a systematic addition of clonidine (150 µg added in the solution bag) in the local anesthetic solution), versus no addition, on the quality of analgesia for labour.

SUMMARY:
In a prospective randomised study involving primiparous women in spontaneous uncomplicated labour with cervical dilatation < 5 cm, epidural analgesia will be given with an initial volume of 20 mL anaesthetic solution, followed by a standardised algorithm of top-up manual injections to achieve analgesia, then by a patient-controlled regimen with 5-mL self-administered boli in addition to a continuous infusion of 5 mL.hr-1. The anaesthetic solution will be levobupivacaine presented in 100-mL bags from the market (0.0625%), in which 10 mL (50 g) of sufentanil will be added, as well as clonidine (150 µg) in one arm. The final concentration of clonidine in this arm will be 1.35 mg.mL-1. Parturients and midwifes assessing pain during labour will be blinded to the design.

DETAILED DESCRIPTION:
We recently compared the analgesic effects of the two presentations of levobupivacaine available on the French market, (0.625 and 1.25 mg.mL-1 in pre-filled bags), both with sufentanil. It appeared that the high concentration was more powerful, however leading in some cases to give doses of levobupivacaine superior to the label's recommendations. This indicates to use the low concentration, with a risk of a poorer efficacy. Our aim is to show that efficacy can be restored with a systematic addition of clonidine, which has documented analgesic properties when administered perispinally.

ELIGIBILITY:
Inclusion Criteria:

* Parturient is 18 years old
* ASA physical status 1 or 2
* Primiparity
* Singleton
* Gestational age is 36 weeks
* Spontaneous labour with cervical dilatation of 5 cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number of required additional epidural boluses, either self-administered or medically given as a rescue | during labour

SECONDARY OUTCOMES:
Spontaneous pain during labour (on VAS) | during labour
Pain at delivery | at delivery
Pain at post-delivery sutures | at post-delivery sutures
Motor block | during labour
Duration of labour | during labour
Obstetrical events (caesarean section, instrumental delivery) | after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Martine Bonnin, MB, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Result] Bazin M, Bonnin M, Storme B, Bolandard F, Vernis L, Lavergne B, Pereira B, Bazin JE, Duale C. Addition of clonidine to a continuous patient-controlled epidural infusion of low-concentration levobupivacaine plus sufentanil in primiparous women during labour. Anaesthesia. 2011 Sep;66(9):769-79. doi: 10.1111/j.1365-2044.2011.06785.x. Epub 2011 Jun 24. PMID 21707560
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/21707560